CLINICAL TRIAL: NCT02088086
Title: Randomized Controlled Trial of BMI Screening: Effects on Obesity, Disparities, and Body Satisfaction
Brief Title: BMI Screening and Reporting in Schools: The Fit Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-07-4472; R01HL120666 (NIH)
Record Dates: First submitted 2014-03-07; First posted 2014-03-14 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Pediatric Obesity; Overweight
Keywords: Pediatric obesity; Overweight; Body mass index; Primary schools; Secondary schools
MeSH Terms: conditions — Pediatric Obesity; Overweight | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BMI screening and reporting (Group 1) (Experimental): For three school years, 3rd-8th grade students will have their heights and weights measured once annually. Additionally, 5th-8th grade students will participate in five fitness assessments. Schools will send BMI reports home to parents.
  Interventions: Behavioral: BMI screening; Behavioral: BMI reporting; Behavioral: Fitness testing
- BMI screening only (Group 2) (Active Comparator): For three school years, 3rd-8th grade students will have their heights and weights measured once annually. Additionally, 5th-8th grade students will participate in five fitness assessments. Schools will NOT send BMI reports home to parents.
  Interventions: Behavioral: BMI screening; Behavioral: Fitness testing
- No BMI screening or reporting (Group 3) (No Intervention): For two school years, 3rd-8th grade students will NOT have their heights and weights measured at school.

INTERVENTIONS:
Behavioral: BMI screening — Students in grades 3-8 will have their heights and weights measured annually at school and their BMIs calculated.
  Arms: BMI screening and reporting (Group 1); BMI screening only (Group 2)
Behavioral: BMI reporting — Schools will send a report home to parents that provides their child's height, weight, and BMI results.
  Arms: BMI screening and reporting (Group 1)
Behavioral: Fitness testing — Students in grades 5-8 will participate in five fitness assessments (curl-ups, sit-ups, push-ups, sit-and-reach, and the PACER test or mile run) annually at school.
  Arms: BMI screening and reporting (Group 1); BMI screening only (Group 2)

SUMMARY:
The Fit Study is a three-year, cluster-randomized controlled trial that will evaluate the impact of school-based body mass index (BMI) screening and reporting on child health. Seventy-nine California schools will be randomized to one of three groups: 1) BMI screening and reporting, 2) BMI screening, and 3) no BMI screening or reporting (control). Investigators will assess the impact of BMI reporting on students' BMI trajectories over three years. Investigators will also assess the impact of BMI screening on weight-based teasing, feelings of stigmatization, and weight-control behaviors among students.

DETAILED DESCRIPTION:
The Fit Study is a three-year, cluster-randomized controlled trial that will evaluate the impact of school-based body mass index (BMI) screening and reporting on childhood obesity and psychosocial outcomes. This study will take place during the 2014-15, 2015-16, and 2016-17 school years. Seventy-nine schools across California will be randomized to one of three groups: 1) BMI screening and reporting, 2) BMI screening, and 3) no BMI screening or reporting (control). Schools randomized to Groups 1 and 2 will conduct height and weight measurements annually with their 3rd-8th grade students. Group 1 and 2 schools will also administer the five fitness assessments (mile run or PACER test, curl-ups, push-ups, trunk lift, and sit and reach) annually with their 5th-8th grade students. In the fall of Years 2 and 3, Group 1 schools will mail a report home to parents with students' results from the previous spring. All 3rd and 4th grade parents will receive a report with BMI results only. Investigators will randomize the parents of 5th-8th grade students to receive a report that provides BMI results only or one that provides BMI results with results from the five fitness assessments. Schools randomized to Group 3 will not conduct height and weight measurements with their students during Years 1 and 2.

Each fall, investigators will administer a survey to 4th-8th grade students from all schools. This survey will assess weight-based teasing, feelings of stigmatization, and weight-control behaviors among students. The student survey will also ask questions about students' experiences having their heights and weights measured at school. During all years, investigators will mail a survey home a subsample of parents to assess parent behaviors related to their child's physical activity and nutrition, as well as parent reactions to the BMI report. Finally, schools will complete a survey in Spring 2017 to assess their nutrition- and physical activity-related policies and programs.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for school districts:

1. District does not report BMI results to caregivers and has no history of doing so
2. District has at least eight schools that meet all of the school-level eligibility criteria

Inclusion criteria for schools:

1. School does not report BMI results to caregivers and has no history of doing so
2. School has an enrollment of 15% to 85% Latino students
3. School has an enrollment of at least 30 students in grades 3 through 8

Inclusion criteria for students: Student is enrolled in 3rd-8th grade

Inclusion criteria for parents: Parent has a child who is enrolled in study

Inclusion criteria for teachers: Teacher measures the heights and weights of students for the study

Exclusion Criteria: None

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36452 (Actual)
Dates: Start 2014-03; Primary Completion 2017-06-15 (Actual); Study Completion 2017-07-15 (Actual)

PRIMARY OUTCOMES:
Change in body mass index (BMI) z-score | Up to 2 years
  Investigators will assess change in BMI z-score over 3 years between students in Group 1 (BMI screening + reporting) and students in Group 2 (BMI screening only). Primary analyses will be limited to students who were overweight (BMI ≥ 85th percentile) at baseline (Spring 2015). Investigators will also compare change in BMI z-score over 3 years between Group 1 students whose parents received the BMI-only report and Group 1 students whose parents received the BMI + fitness report. In both sets of analyses, ethnicity will be used as an effect modifier.

SECONDARY OUTCOMES:
Change in weight-control behaviors | Up to 2 years
  Investigators will compare change in weight-control behaviors (assessed via a survey) between students in Group 3, who did not have their heights and weights measured for 2 school years, and students in Groups 1 and 2, who had their heights and weights measured during those years.
Change in weight-based teasing | Up to 2 years
  Investigators will compare change in experiences of weight-based teasing (assessed via a survey) between students in Group 3, who did not have their heights and weights measured for 2 school years, and students in Groups 1 and 2, who had their heights and weights measured during those years.
Change in body satisfaction | Up to 2 years
  Investigators will compare change in body satisfaction (assessed via a survey) between students in Group 3, who did not have their heights and weights measured for 2 school years, and students in Groups 1 and 2, who had their heights and weights measured during those years.

CONTACTS AND LOCATIONS:
Overall Officials: Kristine A Madsen, MD MPH, Principal Investigator — University of California, Berkeley
Locations (1):
- UC Berkeley School of Public Health, Berkeley, California, United States

REFERENCES:
- [Derived] Madsen KA, Thompson HR, Linchey J, Ritchie LD, Gupta S, Neumark-Sztainer D, Crawford PB, McCulloch CE, Ibarra-Castro A. Effect of School-Based Body Mass Index Reporting in California Public Schools: A Randomized Clinical Trial. JAMA Pediatr. 2021 Mar 1;175(3):251-259. doi: 10.1001/jamapediatrics.2020.4768. PMID 33196797
- [Derived] Thompson HR, Linchey JK, Liu NF, Madsen KA. Parents Recall of, and Reactions to, School-Based BMI Reports. Child Obes. 2019 Dec;15(8):548-554. doi: 10.1089/chi.2019.0061. Epub 2019 Aug 12. PMID 31403338
- [Derived] Thompson HR, Linchey JK, King B, Himes JH, Madsen KA. Accuracy of School Staff-Measured Height and Weight Used for Body Mass Index Screening and Reporting. J Sch Health. 2019 Aug;89(8):629-635. doi: 10.1111/josh.12788. Epub 2019 May 28. PMID 31140199
- [Derived] Madsen KA, Linchey J, Ritchie L, Thompson HR. The Fit Study: Design and rationale for a cluster randomized trial of school-based BMI screening and reporting. Contemp Clin Trials. 2017 Jul;58:40-46. doi: 10.1016/j.cct.2017.05.005. Epub 2017 May 4. PMID 28479218